CLINICAL TRIAL: NCT03696069
Title: Understanding the Treatment Patterns, Healthcare Resource Utilization, Costs of Care, and Clinical Outcomes Among Patients Treated for Advanced Melanoma
Brief Title: A Study is to Understand the Treatment Patterns for Immunotherapy Agents and BRAF/MEK Inhibitors Used in the Treatment of Advanced Melanoma
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8HC
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with immunotherapy and BRAF/MEK inhibitors
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
The goal of the study is to understand the treatment patterns for immunotherapy agents and BRAF/MEK inhibitors used in the treatment of advanced melanoma

ELIGIBILITY:
Inclusion Criteria:

* Patients must have ≥1 medical or pharmacy claim for nivolumab, ipilimumab, pembrolizumab, nivolumab+ipilimumab (on the same day), dabrafenib, vemurafenib, cobimetinib, trametinib, dabrafenib+trametinib (on the same day) and vemurafenib+cobimetinib (on the same day)
* Patients must have ≥6 months of continuous health plan enrollment prior to index date
* Patients must have ≥2 medical claims at least 30 days apart with a diagnosis for melanoma during the study period AND ≥1 diagnosis for melanoma during the baseline period prior to or on the index date

Exclusion Criteria:

* Patients with ≥1 claim for the agents of interest including immunotherapy agents and BRAF/MEK inhibitors between the first diagnosis of metastatic disease and the day prior to the index date will be excluded
* Patients with a claim for acquired immunodeficiency virus (AIDS) anytime during the study period
* Patients under the age of 18 as of index date

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced melanoma treated with immunotherapy and BRAF/MEK inhibitors
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Treatment free interval (TFI) | Approximately 6 months

SECONDARY OUTCOMES:
Overall survival rate | Approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Boston, Massachusetts, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm